CLINICAL TRIAL: NCT00403494
Title: A Phase 2, Multicenter, Multinational, Randomized, Double-blind, Placebo-controlled, Parallel Study of the Effects of Sapropterin Dihydrochloride on Symptomatic Peripheral Arterial Disease
Brief Title: A Phase 2 Study of the Effects of Sapropterin Dihydrochloride on Symptomatic Peripheral Arterial Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PAD-001
Record Dates: First submitted 2006-11-21; First posted 2006-11-23 (Estimated); Results first posted 2021-01-07 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2020-12

CONDITIONS: Intermittent Claudication
Keywords: Intermittent Claudication; IC; Symptomatic Peripheral Arterial Disease; Peripheral Arterial Disease; PAD; 6R-BH4; BH4; sapropterin dihydrochloride; endothelial dysfunction; Nitric Oxide; NO
MeSH Terms: conditions — Intermittent Claudication; Peripheral Arterial Disease | interventions — sapropterin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sapropterin dihydrochloride (Experimental): Subjects receive 400 mg oral sapropterin dihydrochloride twice daily for 24 weeks.
  Interventions: Drug: Sapropterin Dihydrochloride
- Placebo (Placebo Comparator): Subjects receive matching oral Placebo twice daily for 24 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Subjects receive matching oral Placebo twice daily for 24 weeks.
  Arms: Placebo
Drug: Sapropterin Dihydrochloride — Subjects receive 400 mg oral sapropterin dihydrochloride twice daily for 24 weeks.
  Arms: Sapropterin dihydrochloride

SUMMARY:
The purpose of this study is to evaluate whether sapropterin dihydrochloride is safe and effective in the treatment of intermittent claudication (IC) caused by peripheral arterial disease (PAD).

DETAILED DESCRIPTION:
This was a Phase 2, multicenter, multinational, prospective, randomized, double-blind, placebo-controlled, parallel study designed to assess the efficacy and safety of sapropterin dihydrochloride in subjects with intermittent claudication (IC) caused by peripheral arterial disease (PAD). Subjects who met initial screening criteria were monitored criteria and that dosages of permitted concomitant medications were stable.

ELIGIBILITY:
Inclusion Criteria:

* At least 40 years and no more than 80 years old
* A 6-month (or longer) history of walking limitation because of IC, severity of which has not changed in the past 3 months
* Diagnosis of PAD secondary to atherosclerosis, with PAD documented at Screening by one of the following criteria:

  1. Resting ankle-brachial index (ABI) < 0.9 in at least one leg
  2. If resting ABI is 0.9-1.0, minimum post-exercise drop in ABI of at least 25% in at least one leg
  3. If resting ABI is > 1.3 (indicating non-compressible vessels), vascular etiology documented by toe-brachial index (TBI) < 0.7 in at least one leg
* On Gardner graded treadmill protocol, peak walking time (PWT) of at least 1 minute, but no more than 12 minutes
* Variation in PWT between two consecutive screening treadmill tests less than or equal to 25%
* If currently receiving treatment with or taking any of the following, willing and able to discontinue for 30 days before Screening and throughout the entire study (including the follow-up period): phosphodiesterase (PDE) 5 inhibitor (eg, Viagra®, Cialis®, Levitra®, or Revatio™), any PDE 3 inhibitor (eg, cilostazol, milrinone, or vesnarinone), pentoxifylline (Trental®), nitrates, L-arginine, ginkgo biloba, or Heart Bar
* For the approximately 50% of subjects enrolled to receive vitamin C with study drug or placebo, subjects must be willing to discontinue taking vitamin C supplements or a multivitamin containing vitamin C during study.
* Antihypertensive therapy, cholesterol-lowering therapy (eg, statins), and diabetic therapy (if applicable) has been stable for 30 days prior to Screening.
* Has not changed smoking or exercise habits in 30 days prior to randomization and is unlikely to do so during the study period
* Willing and able to provide written, signed informed consent after the nature of the study has been explained and prior to any research-related procedures
* Willing and able to comply with all study-related procedures
* Sexually active subjects must be willing to use an acceptable method of contraception while participating in the study
* Females of childbearing potential must have a negative pregnancy test at Screening and be willing to have additional pregnancy tests during the study

Exclusion Criteria:

* Critical leg ischemia, manifested by pain at rest, ulceration, gangrene, or leg amputation
* Surgical intervention to alleviate symptoms of claudication (eg, vascular reconstruction, sympathectomy) within 6 months or any endovascular interventions or cardiovascular surgery within 3 months
* Walking limited by reasons other than claudication (eg, arthritis, lung disease, exercise-limiting cardiac disease, or skin or foot lesions that limit walking)
* Clinically significant ECG change during or after exercise treadmill test at Screening or Baseline visit(s)
* Myocardial infarction, deep vein thrombosis, or cerebrovascular infarct within 3 months of Screening
* Body mass index > 40 (gross obesity)
* Hypertension at Screening, defined as seated mean resting BP value of > 160 mmHg systolic, > 110 mmHg diastolic, or both
* Hypotension at Screening, defined as seated mean resting BP values of < 100 mmHg systolic or < 55 mmHg diastolic, or as clinically significant symptomatic (orthostatic) hypotension
* Non-atherosclerotic vascular disease (eg, Buerger's disease or popliteal entrapment syndrome)
* Previous treatment with any formulation of BH4
* Known allergy or hypersensitivity to any excipient of 6R-BH4
* Concurrent disease or condition that would interfere with study participation or safety such as bleeding disorders, history of severe gastrointestinal reflux disease, arrhythmia, organ transplant, organ failure, current neoplasm, type 1 diabetes mellitus, or serious neurological disorders (including seizures)
* Previous treatment with gene therapy or other vascular endothelial growth factor (VEGF)-related treatment
* Any severe co-morbid condition that would limit life expectancy to less than 6 months
* Serum creatinine > 2.0 mg/dL or hepatic enzyme levels more than 2 times the upper limit of normal
* Concomitant treatment with levodopa
* Requirement for concomitant treatment with any drug known to inhibit folate metabolism (eg, methotrexate)
* Use of any investigational product or device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments
* Pregnant or breastfeeding at Screening or planning to become pregnant (subject or partner) at any time during the study

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2006-12; Primary Completion 2008-11 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Don Nwose, MD, Study Director — BioMarin Pharmaceutical
Locations (20):
- United States (17):
  - Scottsdale, Arizona
  - Sacramento, California
  - San Diego, California
  - Santa Ana, California
  - Santa Rosa, California
  - Clearwater, Florida
  - Jacksonville, Florida
  - Conyers, Georgia
  - Indianapolis, Indiana
  - Auburn, Maine
  - Charlotte, North Carolina
  - Portland, Oregon
  - Knoxville, Tennessee
  - Dallas, Texas
  - San Antonio, Texas
  - Norfolk, Virginia
  - Richmond, Virginia
- Argentina (3):
  - Buenos Aires
  - Corrientes
  - Santa Fe

REFERENCES:
- See also: BioMarin Pharmaceutical Inc. website — http://www.bmrn.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a multicenter, multinational study. 31 principal investigators (PIs) enrolled subjects at 10 sites in Argentina sites and 21 sites in the United States (US). A total of 190 patients were recruited with 96 subjects randomized to Sapropterin dihydrichloride and 94 to Placebo. 65 subjects were in Argentina - (32 Sapropterin dihydrochloride, 33 Placebo), and 125 subjects in the US - (64 Sapropterin dihydrochloride, 61 Placebo)
Groups:
- Placebo: Subjects receive matching oral Placebo twice daily for 24 week.
Period: Overall Study
Arm/Group | Sapropterin Dihydrochloride | Placebo
Started | 96 | 94
Intent to Treat (All subjects who were randomized, received 1 dose of study drug and had at least 1 post-baseline treadmill assessment,) | 87 | 83
Per-protocol (The Per-protocol population will exclude subjects with major protocol deviations or noncompliance of study procedures. Including subjects that did not complete week 24 treadmill test, took less than 80% of the randomized study drug, and/or experienced any acute confounding events preventing them from taking proper treadmill tests.) | 69 | 69
Safety Population (Of the 188 patients (96 randomized to study drug and 94 to placebo.) 2 subjects randomized to receive placebo, received at least 1 dose of study drug and were included in the study drug group. 1 participant from each group was excluded from the safety analysis because they did not have at least 1 post-Baseline safety assessment.) | 97 | 91
Completed | 81 | 80
Not Completed | 15 | 14
Not completed — Adverse Event | 10 | 8
Not completed — Withdrew Consent | 3 | 2
Not completed — Inappropriately enrolled | 0 | 1
Not completed — Lost to Follow-up | 0 | 2
Not completed — Protocol noncompliance | 0 | 1
Not completed — Death | 1 | 0
Not completed — Sponsor Request | 1 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population
Groups:
- Total: Total of all reporting groups
Arm/Group | Sapropterin Dihydrochloride | Placebo | Total
Number analyzed (Participants) | 87 | 83 | 170
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (8.9) | 66.6 (7.0) | 67.3 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 45
  Male | 65 | 60 | 125
Age [Count of Participants; unit: Participants]
  < 65 years | 28 | 35 | 63
  >= 65 years | 59 | 48 | 107
  >= 75 years | 25 | 10 | 35
Race [Count of Participants; unit: Participants]
  White | 80 | 75 | 155
  Black/African American | 5 | 7 | 12
  Other | 2 | 0 | 2
  Asian | 0 | 1 | 1
Ethnicity [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 58 | 52 | 110
  Hispanic or Latino | 29 | 31 | 60
Country of Study Site [Count of Participants; unit: Participants]
  United States | 60 | 53 | 113
  Argentina | 27 | 30 | 57
With/Without Vitamin C [Count of Participants; unit: Participants] — Vitamin C (500 mg/2X per day orally) was added to the study drug dose for the last 50% of enrolled patients to assess impact on sapropterin dihydrochloride absorption.
  Participants
    Without Vitamin C | 41 | 39 | 80
    With Vitamin C | 46 | 44 | 90

OUTCOME MEASURES:

1. Primary Outcome: Change in Peak Walking Time (PWT) From Baseline
Description: This is to assess the effect of oral sapropterin dihydrochloride versus placebo on peak walking time (PWT) in subjects with intermittent claudication (IC) caused by peripheral arterial disease (PAD).
Time Frame: Baseline and up to Week 24
Population: Intent-To-Treat Population consisting of all subjects who were randomized, received 1 dose of study drug and had at least 1 post-baselline treadmill test.
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Sapropterin Dihydrochloride: Intent to Treat Population. Subjects receive 400 mg oral sapropterin dihydrochloride twice daily for 24 weeks
- Placebo: Intent to Treat Population. Subjects receive matching oral Placebo twice daily for 24 weeks.
Arm/Group | Sapropterin Dihydrochloride | Placebo
Number analyzed (Participants) | 87 | 83
minutes
  Baseline | 5.394 (2.803) | 5.712 (2.876)
  Change from Baseline to Week 24: number analyzed (Participants) | 82 | 80
  Change from Baseline to Week 24 | 1.121 (2.775) | 1.493 (2.597)
Statistical Analysis 1: Comparison: Sapropterin Dihydrochloride vs Placebo; Test type: Superiority — PWT was transformed to the log ratio at Week 24:Baseline for statistical analysis; p = 0.727, t-test, 2 sided; Mean Difference (Final Values) = -0.021, 95% CI 2-sided [-0.138 to 0.097], Standard Deviation 0.379 — Mean difference represents the difference of the means of the natural log-transformed ratios between the 2 treatment groups

2. Primary Outcome: Number of Subjects With Adverse Events (AEs)
Description: Adverse events were described and summarized with focus on treatment- emergent events (TEAEs). A TEAE was defined as any AE that presented , increased in frequency or worsened in severity following initiation of study drug administration. If the onset of an AE was missing then the AE was considered treatment emergent. Drug-related AEs are AEs classified by the investigator as possibly or probably related to study drug.
Time Frame: Up to 24-weeks
Population: Of the 188 patients (96 randomized to study drug and 94 to placebo.) 2 subjects randomized to receive placebo, received at least 1 dose of study drug and were included in the study drug group. 1 participant from each group was excluded from the safety analysis because they did not have at least 1 post-Baseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Sapropterin Dihydrochloride | Placebo
Number analyzed (Participants) | 97 | 91
Participants
  Any AEs | 84 | 66
  Study Drug-related AEs | 29 | 30
  Any SAEs | 14 | 11
  Study-Drug-related SAEs | 0 | 1
  Any AEs leading to Study Withdrawal | 11 | 7
  Study Drug-related AEs leading to Study WIthdrawal | 4 | 5
  Any SAEs Leading to Study Withdrawal | 4 | 1
  Study Drug-related SAEs Leading to Study Withdrawal | 0 | 1
  Deaths | 1 | 0

3. Secondary Outcome: Change in Claudication Onset Time (COT) From Baseline
Description: Time, in minutes, when the subject first begins to experience claudication symptoms, regardless of whether this is manifested as muscle pain, ache, cramp, numbness or fatigue.
Time Frame: Baseline and up to Week 24
Population: Intent-To-Treat Population
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sapropterin Dihydrochloride | Placebo
Number analyzed (Participants) | 87 | 83
minutes
  Baseline | 2.159 (1.611) | 2.313 (1.689)
  Change from Baseline to Week 24: number analyzed (Participants) | 80 | 78
  Change from Baseline to Week 24 | 0.903 (1.900) | 1.015 (1.902)

4. Other Pre Specified Outcome: Change in Peak Walking Time From Baseline With and Without Vitamin C
Description: The first 50% of subjects enrolled in the study were randomized to receive sapropterin dihydrochloride at 400 mg BID or oral placebo BID alone (without vitamin C). When approximately 50% enrollment was met, 1000 mg/day vitamin C was added to the dose regimen of newly enrolled subjects in both sapropterin dihydrochloride and placebo treatment groups given orally in two divided doses of 500 mg with study drug.
Time Frame: Baseline up to 24 weeks
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Sapropterin Dihydrochloride | Placebo
Number analyzed (Participants) | 87 | 83
minutes
  Baseline without vitamin C: number analyzed (Participants) | 41 | 39
  Baseline without vitamin C | 4.776 (2.650) | 5.201 (2.781)
  Change from Baseline week 24; without vitamin C: number analyzed (Participants) | 37 | 37
  Change from Baseline week 24; without vitamin C | 0.264 (2.064) | 0.607 (2.166)
  Baseline with vitamin C: number analyzed (Participants) | 46 | 44
  Baseline with vitamin C | 5.944 (2.849) | 6.164 (2.914)
  Change from Baseline week 24; with vitamin C: number analyzed (Participants) | 45 | 43
  Change from Baseline week 24; with vitamin C | 1.826 (3.093) | 2.255 (2.716)

ADVERSE EVENTS:
Time Frame: Up to 25 Weeks
Description: Of the 188 patients (96 randomized to study drug and 94 to placebo.) 2 subjects randomized to receive placebo, received at least 1 dose of study drug and were included in the study drug group. 1 participant from each group was excluded from the safety analysis because they did not have at least 1 post-Baseline safety assessment.
Arm/Group | Sapropterin Dihydrochloride | Placebo
All-Cause Mortality (participants affected / at risk) | 1/97 | 0/91
Serious Adverse Events (participants affected / at risk) | 14/97 | 11/91
Other Adverse Events (participants affected / at risk) | 84/97 | 66/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sapropterin Dihydrochloride (N=97) | Placebo (N=91)
Acute coronary syndrome (Vascular disorders) | 0 | 1
Angina unstable (Vascular disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 1 | 0
Cerebrovascular accident (Vascular disorders) | 1 | 0
Coronary artery disease (Vascular disorders) | 1 | 0
Gastric haemorrhage (Vascular disorders) | 0 | 1
Ischaemic limb pain (Vascular disorders) | 1 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 1
Renal artery stenosis (Vascular disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Retroperitoneal neoplasm (Gastrointestinal disorders) | 1 | 0
Electrocardiogram abnormal (Investigations) | 0 | 1
Prostate examination abnormal (Investigations) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Death (General disorders) | 1 | 0 — Term as reported. It was noted patient was found dead in home. No autopsy was done.
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Alcoholism (Psychiatric disorders) | 0 | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sapropterin Dihydrochloride (N=97) | Placebo (N=91)
Diarrhoea (Gastrointestinal disorders) | 4 | 7
Nausea (Gastrointestinal disorders) | 5 | 4
Pharmaceutical product complaint (General disorders) | 4 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 1
Nasopharyngitis (Infections and infestations) | 6 | 3
Headache (Nervous system disorders) | 4 | 5
Hypotension (Vascular disorders) | 8 | 0
Intermittent claudication (Vascular disorders) | 6 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 3
Abdominal Pain Upper (Gastrointestinal disorders) | 4 | 1
Fatigue (General disorders) | 4 | 4
Hypertension (Vascular disorders) | 4 | 4
Oedema peripheral (General disorders) | 4 | 4
Upper respiratory tract infection (Infections and infestations) | 4 | 3
Bronchitis (Infections and infestations) | 3 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 1
Insomnia (Nervous system disorders) | 3 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 3
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 3 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3 | 0
Urinary tract infection (Infections and infestations) | 3 | 3
Flatulence (Gastrointestinal disorders) | 2 | 5
Dyspepsia (Gastrointestinal disorders) | 0 | 5
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days